CLINICAL TRIAL: NCT02849197
Title: Comparative Analysis of the Same technique-the Same Surgeon Approach in the Surgical Treatment of Pilonidal Sinus Disease: A Retrospective Cohort Study
Brief Title: Study on Surgical Treatment of Pilonidal Sinus Disease
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Mustafa Hasbahceci, associate professor, Bezmialem Vakif University
Other Study IDs: PilonidalSinus-EK/MH
Record Dates: First submitted 2016-07-20; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Pilonidal Sinus
Keywords: pilonidal sinus; complication; recurrence
MeSH Terms: conditions — Pilonidal Sinus; Recurrence | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Primary Closure: Patients with pilonidal sinus disease treated with surgery for pilonidal sinus disease.
  Technique: primary closure. Technical details: An elliptical incision was made, and the excision included sinus openings at the median line and extended down to the pre-sacral fascia. One suction drain was placed in the wound cavity. Subcutaneous tissue was approximated with interrupted 2-0 absorbable suture, and skin was closed with interrupted 2-0 silk suture.
  Interventions: Procedure: surgery for pilonidal sinus disease
- Limberg Flap Technique: Patients with pilonidal sinus disease treated with surgery for pilonidal sinus disease.
  Technique: Limberg Flap Technique. Technical details: A rhomboid incision was made as to include all sinus openings, and an excision was made down to the pre-sacral fascia. A bisector drawn in the rhombohedron was extended laterally to a length similar to that of a corner of the rhombohedron. Then, the flap was prepared by removing gluteal muscle with its fascia. One suction drain was placed at the wound cavity. The base of the flap was approximated with the presacral fascia at the excised area with interrupted 2-0 absorbable sutures. Subcutaneous tissue was approximated with interrupted 2-0 absorbable sutures, and the skin was closed with interrupted 3-0 prolene suture.
  Interventions: Procedure: surgery for pilonidal sinus disease
- Modified Limberg Technique: Patients with pilonidal sinus disease treated with surgery for pilonidal sinus disease.
  Technique: Modified Limberg Flap Technique. Technical details: As in Limberg flap technique, a rhomboid incision was made. Upper and lower corners of the excision were lateralized 2 cm away from the midline in order to keep the suturing line at the inferior from overlapping the midline. An excision was made down to the pre-sacral fascia. One suction drain was placed at the wound cavity, and the base of the flap was approximated with the pre-sacral fascia at the excised area with interrupted 2-0 absorbable sutures. Subcutaneous tissue was approximated with interrupted 2-0 absorbable suture, and the skin was closed with 3-0 prolene.
  Interventions: Procedure: surgery for pilonidal sinus disease

INTERVENTIONS:
Procedure: surgery for pilonidal sinus disease — surgical treatment of pilonidal sinus disease via primary closure, Limberg flap0 technique and Modified Limberg flap technique.

SUMMARY:
Comparison of limited excision-primary closure, Limberg, and modified Limberg flap techniques for the surgical treatment of pilonidal sinus disease, each performed by a separate surgeon, in terms of postoperative outcomes and recurrence rates.

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) is a common chronic disease that generally affects young adults below the age of 45. It is most commonly observed at the inter-gluteal region, though it may also affect other sites like the umbilicus and the inter-digital area, particularly among in barbers. The disease was long thought to be either congenital or acquired; although in recent years it has been more widely viewed as an acquired disease. The etiology of PSD is not fully understood, however, the most important cause is believed to be fallen hairs accumulating within skin folds and implanting within the skin. The skin becomes more prone to maceration, sweating and bacterial contamination, which facilitates implantation of fallen hairs, creating the necessary conditions for development of the disease. Although PSD is a benign disease, it produces symptoms such as pain and discharge, which adversely affect patient quality of life.

There are many approaches for treatment of the disease, including several surgical methods such as limited or large excision, primary closure, or flap techniques, and many other non-surgical methods. However, no consensus has been reached regarding the ideal treatment method. An ideal surgical treatment reduces recurrence and complication rates, and allows for minimal hospitalization and rapid return to daily activities. Among patients treated using the limited excision and primary closure method, the presence of a natal cleft is associated with higher morbidity, resulting in recurrence rates of 7-42%. For techniques that use the flap approach, this rate decreases to 0-3%. In patients undergoing the Rhomboid excision and Limberg flap techniques, which require a larger surgical area compared to the limited excision and primary closure methods, complication rates are lower, and length of hospital-stay and time to return to work are reduced. However, using the classical Limberg flap technique, maceration and scar formation due to sutures in the inter-gluteal sulcus, and the accumulation of hair at the midline may result in recurrence. Application of a modified Limberg technique that includes lateralization of the middle line can help reduce wound complications and recurrence rates. Several publications report contradicting results regarding surgical outcomes using the same technique, which may be attributable to differences in practice between surgeons. Therefore, it can be logical to explore the superiority of any type of surgical technique performed by the same surgeon for the surgical treatment of pilonidal sinus disease.

ELIGIBILITY:
Inclusion Criteria:

* patients who were diagnosed with pilonidal sinus disease and who underwent surgical treatment in a governmental hospital between January 2011 and June 2015

Exclusion Criteria:

* patients with incomplete personal and medical data and who could not be contacted by direct interview or by telephone

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 1082 patients who were diagnosed with pilonidal sinüs disease and who underwent surgical treatment in a governmental hospital between January 2011 and June 2015.
Sampling Method: Non-Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion at an average of 36 months

CONTACTS AND LOCATIONS:
Overall Officials: mustafa hasbahceci, assoc. prof., Principal Investigator — Bezmialem Vakif University

IPD SHARING:
Plan to Share IPD: No